CLINICAL TRIAL: NCT05632471
Title: The Effect of Web-Based Education Given to Parents on Children's İnternet Gaming Disorder
Brief Title: The Effect of Web-based Education Given to Parents on Children's Internet Gaming Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Meryem MUTLU, Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMUTLU
Record Dates: First submitted 2022-11-06; First posted 2022-11-30 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Internet Gaming Disorder
Keywords: Internet Gaming Disorder; Parents; Prevention methods; Child; Web-Based Education
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web-based training for parents in the intervention group (Experimental): Parents were given "I know digital games" training with 10 videos from the website.
  Interventions: Behavioral: web-based "I know digital games" training for intervation grup
- parents in the control group (Other): No intervention was applied to the parents in the control group.
  Interventions: Other: The control group was not trained

INTERVENTIONS:
Behavioral: web-based "I know digital games" training for intervation grup — "I know digital games" training consisting of 10 web-based videos
  Arms: web-based training for parents in the intervention group
Other: The control group was not trained — The control group was not trained
  Arms: parents in the control group

SUMMARY:
Internet Gaming Disorder (IOB) is an important problem that is increasingly prevalent all over the world and can be prevented before it develops. This research is a single-blind, randomized controlled experimental study to evaluate the effect of Internet-based education given to parents on children's Internet gaming disorder. 96 children and their parents studying in the central districts of a province and at risk for the development of IOBB were divided into intervention (48) and control groups (48) according to the randomization list. The "I know digital games" training consisting of three modules and 10 videos was given to the intervention group via the website prepared by the researchers, and no intervention was made to the control group. The research data were collected at three different times using the "Internet Gaming Disorder Scale Short Form" (İOOBÖ9-SF) and the forms developed by the researchers. In the analysis of data; descriptive statistics, Chi-square, Mann Whitney U test, and repeated measures ANOVA were used. Before the analysis, eight missing data in the control group were estimated with regression estimation models from intent to treat protocols. Statistical significance level p ≤0.05 was taken in all analyzes. Parents and children in the intervention and control groups were similar in terms of sociodemographic characteristics and playing characteristics (p>0.05). It would be beneficial to involve parents in the interventions that nurses will make for primary school children in order to prevent IOB.

ELIGIBILITY:
Inclusion Criteria:

* For kids

  * To have a score between 25-36 from IOOBÖ9-SF [69]
  * Willingness to participate in the study,
  * No communication barrier,
  * Being educated in high socioeconomic level schools,
  * Not having a psychiatric diagnosis and/or not using psychiatric medication
* for parents

  * Your child's score between 25-36 on IOOBÖ9-SF,
  * Willingness to participate in the study,
  * No communication barrier,
  * Having at least one tablet/smartphone/computer and being able to use these devices,
  * Having mobile or home internet,
  * Being literate,
  * The parent who will participate in the study does not have a psychiatric diagnosis and/or uses psychiatric medication.

Exclusion Criteria:

* For kids

  * Having received 25 points below or 36 points above IOOBÖ9-SF
  * Not being willing to participate in the study,
  * Having a communication barrier (not being able to speak or understand Turkish…),
  * Having a psychiatric diagnosis and/or using psychiatric medication
* for parents

  * Your child's score below 25 or above 36 on OOOBÖ9-SF
  * Not being willing to participate in the study,
  * Having a communication barrier (not being able to speak or understand Turkish…)
  * Not having at least one tablet/smartphone/computer,
  * Not having mobile or home internet,
  * Being illiterate,
  * The parent who will participate in the study does not have a psychiatric diagnosis and/or uses psychiatric medication.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Internet Gaming Disorder Scale Short Form (IGDS9-SF) score | 4 months
  An increase in the scale scores means that the problematic behavior increases. (Min:9; Max:36)

SECONDARY OUTCOMES:
Parents' knowledge points on digital games | 4 months
  Evaluation of parents' knowledge scores about digital games
Families' Knowledge, Behavior and Problems Related to Digital Games Evaluation Form scores | 4 months
  Evaluation of the scores obtained by parents from the form in the dimensions of "controlling their children's digital games", "protecting them from the harms of digital games", "limiting their digital games", "forcefully controlling (punishing) digital games", "guiding digital games".
Problems that parents have with their children due to digital games | 4 months
  Evaluation of the problems parents experience with their children due to digital games
children's digital gaming time | 4 months
  Evaluation of children's digital game playing time

CONTACTS AND LOCATIONS:
Overall Officials: Sümbüle Köksoy Vayısoğlu, Study Director — Mersin University Faculty of Nursing
Locations (1):
- Meryem MUTLU SAYIN, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Will be shared after the completion of the research reports.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It can be used for two years after the research reports are uploaded.
Access Criteria: To be doing research on digital addictions.